CLINICAL TRIAL: NCT01025791
Title: A Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8266
Brief Title: A Single Dose Study of MK-8266 (MK-8266-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 8266-001; MK-8266-001 (Other: Merck protocol number); 2009_700 (Other: Telerx ID); 2009-015774-36 (EudraCT Number)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Panel A, Healthy Male Participants, Sequence 1 (Experimental): MK-8266 in Period 1: 0.1 mg/ Period 2: 0.2 mg/ Period 3: placebo/ Period 4: 1.0 mg/ Period 5: 1.0 mg dose followed in 6 hours by a 0.8 mg dose.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel A, Healthy Male Participants, Sequence 2 (Experimental): MK-8266 in Period 1: 0.1 mg/ Period 2: 0.2 mg/ Period 3: 0.5 mg/ Period 4: placebo/ Period 5: 1.0 mg dose followed in 6 hours by a 0.8 mg dose.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel A, Healthy Male Participants, Sequence 3 (Experimental): MK-8266 in Period 1: 0.1 mg/ Period 2: placebo/ Period 3: 0.5/ Period 4: 1.0 mg/ Period 5: placebo.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel A, Healthy Male Participants, Sequence 4 (Experimental): MK-8266 in Period 1: placebo/ Period 2: 0.2 mg/ Period 3: 0.5 mg/ Period 4: 1.0 mg/ Period 5: 1.0 mg dose followed in 6 hours by a 0.8 mg dose.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel B, Healthy Male Participants, Sequence 1 (Experimental): MK-8266 in Period 1: 0.4 mg/ Period 2: 1.2 mg/ Period 3: placebo/ Period 4: 0.4 mg fed/ Period 5: na.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel B, Healthy Male Participants, Sequence 2 (Experimental): MK-8266 in Period 1: 0.4 mg/ Period 2: placebo/ Period 3: 1.2 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 0.4 mg fed/ Period 5: na.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel B, Healthy Male Participants, Sequence 3 (Experimental): MK-8266 in Period 1: 0.4 mg/ Period 2: 1.2 mg/ Period 3: 1.2 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 0.4 mg fed/ Period 5: na.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg
- Panel B, Healthy Male Participants, Sequence 4 (Experimental): MK-8266 in Period 1: placebo/ Period 2: 1.2 mg/ Period 3: 1.2 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: placebo/ Period 5: na.
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel C, Mild/Moderate Hypertension, Sequence 1 (Experimental): Period 1: placebo/ Period 2 1.2 mg dose followed in 8 hours by a 1.0 mg dose/ Period 3: 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg
- Panel C, Mild/Moderate Hypertension, Sequence 2 (Experimental): Period 1: placebo/ Period 2 1.2 mg dose followed in 8 hours by a 1.0 mg dose/ Period 3: 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: placebo/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel C, Mild/Moderate Hypertension, Sequence 3 (Experimental): Period 1: 1.0 mg dose followed in 8 hours by a 0.8 mg dose/ Period 2 placebo/ Period 3: 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel C, Mild/Moderate Hypertension, Sequence 4 (Experimental): Period 1: 1.0 mg dose followed in 8 hours by a 0.8 mg dose/ Period 2: placebo/ Period 3: 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: placebo/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo
- Panel C, Mild/Moderate Hypertension, Sequence 5 (Experimental): Period 1: 1.0 mg dose followed in 8 hours by a 0.8 mg dose/ Period 2: 1.2 mg dose followed in 8 hours by a 1.0 mg dose// Period 3: placebo/ Period 4: 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg
- Panel C, Mild/Moderate Hypertension, Sequence 6 (Placebo Comparator): Period 1: 1.0 mg dose followed in 8 hours by a 0.8 mg dose/ Period 2: 1.2 mg dose followed in 8 hours by a 1.0 mg dose// Period 3: placebo/ Period 4: placebo/ Period 5: na
  Interventions: Drug: MK-8266 0.1 mg; Drug: MK-8266 1.0 mg; Drug: Placebo

INTERVENTIONS:
Drug: MK-8266 0.1 mg — Single oral doses of 0.1 to 1.2 mg of MK-8266 in 0.1 capsule form. Participants will fast for 8 hours prior to dosing. There will be at least a 7- day washout period between doses for any given participant. Some participants will receive study drug with food.
  Other Names: MK-8266
Drug: MK-8266 1.0 mg — MK-8266 1.0 mg oral capsule. Participants will fast for 8 hours prior to dosing. There will be at least a 7- day washout period between doses for any given participant.
Drug: Placebo — Placebo to match MK-8266 0.1 or 1.0 mg. Participants will fast for 8 hours prior to dosing. There will be at least a 7- day washout period between doses for any given participant.
  Arms: Panel A, Healthy Male Participants, Sequence 1; Panel A, Healthy Male Participants, Sequence 2; Panel A, Healthy Male Participants, Sequence 3; Panel A, Healthy Male Participants, Sequence 4; Panel B, Healthy Male Participants, Sequence 1; Panel B, Healthy Male Participants, Sequence 2; Panel B, Healthy Male Participants, Sequence 4; Panel C, Mild/Moderate Hypertension, Sequence 2; Panel C, Mild/Moderate Hypertension, Sequence 3; Panel C, Mild/Moderate Hypertension, Sequence 4; Panel C, Mild/Moderate Hypertension, Sequence 6

SUMMARY:
A three panel study, to determine if MK-8266 given as a single dose is sufficiently safe and well tolerated. Panel A and B will consist of healthy young males and Panel C will consist of subjects with mild to moderate hypertension. The primary hypotheses for the study are that MK-8266 given as single doses is sufficiently safe and well tolerated to permit continued clinical investigation in healthy young male volunteers and male participants with mild-to-moderate hypertension and that in males with mild to moderate hypertension, at a single oral dose of MK-8266 that is sufficiently safe and well-tolerated, postdose mean time-weighted average across 24 hours of aortic augmentation index (TWA0-12hrs AIx) is reduced compared to placebo. A mean decrease of ≥ 5 percentage points is considered clinically meaningful.

DETAILED DESCRIPTION:
Three panels, each consisting of either 8 or 9 participants (8 healthy young males in Panel A and Panel B; and 9 participants with mild to moderate hypertension in Panel C) will be randomized to receive either MK-8266 or matching placebo in either a 6:2 ratio (Panel A and Panel B) or 6:3 ratio (Panel C), respectively, in up to 5 treatment (1 to 5) periods in Panel A and up to 4 treatment (1 to 4) periods in Panel B and Panel C. In all panels, doses will be escalated in a rising, fixed sequence. Some participants took study drug after fasting and some with food.

ELIGIBILITY:
Inclusion Criteria:

* For Panel A and B Participant is a healthy male between 18 to 45 years of age. For Panel C Participant is a male with essential hypertension between 18 to 55 years of age
* A non-smoker

Exclusion Criteria:

* Has a history of stroke, chronic seizure or major neurological disorder
* Has a disability that can interfere with rising from a sitting position to the standing position
* Has a personal of family history of bleeding or clotting disorders
* Has a history of cancer
* Is unable to refrain from or anticipates the use of any prescription or nonprescription drug during the study
* Consumes excessive amounts of caffeine or alcohol
* Has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2010-05-14 (Actual); Study Completion 2010-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 2 clinical study sites in Germany and in Belgium.
Pre-assignment Details: For Panel A, 5 treatment periods were planned in this study. For Panels B and C, only 4 treatment periods were planned.
Period: Period 1
Arm/Group | Panel A, Healthy Male Participants, Sequence 1 | Panel A, Healthy Male Participants, Sequence 2 | Panel A, Healthy Male Participants, Sequence 3 | Panel A, Healthy Male Participants, Sequence 4 | Panel B, Healthy Male Participants, Sequence 1 | Panel B, Healthy Male Participants, Sequence 2 | Panel B, Healthy Male Participants, Sequence 3 | Panel B, Healthy Male Participants, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 1 | Panel C, Mild/Moderate Hypertension, Sequence 2 | Panel C, Mild/Moderate Hypertension, Sequence 3 | Panel C, Mild/Moderate Hypertension, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 5 | Panel C, Mild/Moderate Hypertension, Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Panel A, Healthy Male Participants, Sequence 1 | Panel A, Healthy Male Participants, Sequence 2 | Panel A, Healthy Male Participants, Sequence 3 | Panel A, Healthy Male Participants, Sequence 4 | Panel B, Healthy Male Participants, Sequence 1 | Panel B, Healthy Male Participants, Sequence 2 | Panel B, Healthy Male Participants, Sequence 3 | Panel B, Healthy Male Participants, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 1 | Panel C, Mild/Moderate Hypertension, Sequence 2 | Panel C, Mild/Moderate Hypertension, Sequence 3 | Panel C, Mild/Moderate Hypertension, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 5 | Panel C, Mild/Moderate Hypertension, Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Panel A, Healthy Male Participants, Sequence 1 | Panel A, Healthy Male Participants, Sequence 2 | Panel A, Healthy Male Participants, Sequence 3 | Panel A, Healthy Male Participants, Sequence 4 | Panel B, Healthy Male Participants, Sequence 1 | Panel B, Healthy Male Participants, Sequence 2 | Panel B, Healthy Male Participants, Sequence 3 | Panel B, Healthy Male Participants, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 1 | Panel C, Mild/Moderate Hypertension, Sequence 2 | Panel C, Mild/Moderate Hypertension, Sequence 3 | Panel C, Mild/Moderate Hypertension, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 5 | Panel C, Mild/Moderate Hypertension, Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Panel A, Healthy Male Participants, Sequence 1 | Panel A, Healthy Male Participants, Sequence 2 | Panel A, Healthy Male Participants, Sequence 3 | Panel A, Healthy Male Participants, Sequence 4 | Panel B, Healthy Male Participants, Sequence 1 | Panel B, Healthy Male Participants, Sequence 2 | Panel B, Healthy Male Participants, Sequence 3 | Panel B, Healthy Male Participants, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 1 | Panel C, Mild/Moderate Hypertension, Sequence 2 | Panel C, Mild/Moderate Hypertension, Sequence 3 | Panel C, Mild/Moderate Hypertension, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 5 | Panel C, Mild/Moderate Hypertension, Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Panel A, Healthy Male Participants, Sequence 1 | Panel A, Healthy Male Participants, Sequence 2 | Panel A, Healthy Male Participants, Sequence 3 | Panel A, Healthy Male Participants, Sequence 4 | Panel B, Healthy Male Participants, Sequence 1 | Panel B, Healthy Male Participants, Sequence 2 | Panel B, Healthy Male Participants, Sequence 3 | Panel B, Healthy Male Participants, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 1 | Panel C, Mild/Moderate Hypertension, Sequence 2 | Panel C, Mild/Moderate Hypertension, Sequence 3 | Panel C, Mild/Moderate Hypertension, Sequence 4 | Panel C, Mild/Moderate Hypertension, Sequence 5 | Panel C, Mild/Moderate Hypertension, Sequence 6
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel A MK-8266 (Healthy Males): MK-8266 single dose or placebo matching MK-8266 in healthy male participants in Period 1: 0.1 mg/ Period 2: 0.2 mg/ Period 3: 0.5 mg/ Period 4: 1.0 mg/ Period 5: 1.0 mg dose followed in 6 hours by a 0.8 mg dose.
- Panel B MK-8266 (Healthy Males): MK-8266 single dose or placebo matching MK-8266 in healthy male participants in Periods 1: 0.4 mg/ Period 2: 1.2 mg/ Period 3: 1.2 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 0.4 mg fed/ Period 5: na.
- Panel C MK-8266 (Mild/Mod. Hypertension): MK-8266 single dose or placebo matching MK-8266 (Mild/Mod. Hypertension) in Period 1: 1.0 mg dose followed in 8 hours by a 0.8 mg dose/ Period 2: 1.2 mg dose followed in 8 hours by a 1.0 mg dose/ Period 3: 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose/ Period 4: 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose/ Period 5: na
- Total: Total of all reporting groups
Arm/Group | Panel A MK-8266 (Healthy Males) | Panel B MK-8266 (Healthy Males) | Panel C MK-8266 (Mild/Mod. Hypertension) | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (8.1) | 27.3 (5.4) | 47.3 (3.9) | 36.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Participants in Arms/Groups in which MK-8266 or placebo was administered in more than one period were counted separately for each period.
Time Frame: Up to 14 days after administration of last dose of study drug in each study period (Up to 43 Days)
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A MK-8266 0.1 mg (Healthy Males): MK-8266 single 0.1 mg dose in healthy male participants
- Panel A MK-8266 0.2 mg (Healthy Males): MK-8266 single 0.2 mg dose in healthy male participants
- Panel A MK-8266 0.5 mg (Healthy Males): MK-8266 single 0.5 mg dose in healthy male participants
- Panel A MK-8266 1.0 mg (Healthy Males): MK-8266 single 1.0 mg dose in healthy male participants
- Panel A MK-8266 1.0/0.8 mg (Healthy Males): MK-8266 single 1.0 mg dose followed in 6 hours by a 0.8 mg dose in healthy male participants
- Panel B MK-8266 0.4 mg (Healthy Males): MK-8266 single dose 0.4 mg in healthy male participants
- Panel B MK-8266 1.2 mg (Healthy Males): MK- 8266 single dose 1.2 mg in healthy male participants
- Panel B MK-8266 1.2/0.6 mg (Healthy Males): MK-8266 single 1.2 mg followed in 6 hours by a 0.6 mg dose in healthy male
- Panel B MK-8266 0.4 mg Fed (Healthy Males): MK-8266 single 0.4 mg dose in healthy male participants, fed.
- Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension): MK-8266 single 1.0 mg dose followed in 8 hours by a 0.8 mg dose in participants with mild/mod. hypertension
- Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension): MK-8266 single 1.2 mg dose followed in 8 hours by a 1.0 mg dose in participants with mild/mod. hypertension
- Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension): MK-8266 single 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose in participants with mild/mod. hypertension
- Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension): MK-8266 single 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose in participants with mild/mod. hypertension
- Pooled Placebo (Panels A, B, C): Placebo matching MK-8266.
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) | Pooled Placebo (Panels A, B, C)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 23
Participants | 2 | 3 | 5 | 2 | 3 | 1 | 4 | 3 | 2 | 3 | 4 | 6 | 3 | 10

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 1
Time Frame: Up to 43 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) | Pooled Placebo (Panels A, B, C)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Aortic Augmentation Index - Time-Weighted Average 0-24 Hours
Description: Central ascending aortic blood pressure augmentation index (AIx) is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. AIx can be measured non-invasively by radial tonometry using aplanation tonometry of radial artery with the SphygmoCor Pulse Wave Analysis System Guide (SphygmoCor system). AIx was performed at prestudy to ensure an adequate waveform can be obtained. At each time point, a minimum of 2 AIx were completed in an attempt to obtain 2 acceptable quality assessments. A time weighted average was calculated. AIx was adjusted for heart rate. A decrease in the AIx of ≥5 percentage is considered clinically meaningful. Participants in Arms/Groups in which MK-8266 or placebo was administered in more than one period were counted separately for each period. The 12-hour measurement was not collected (per protocol) in all periods of Panels A and B.
Time Frame: Predose, 1.5, 3, 12, and 24 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that their data likely exhibited the effects of treatment. Panel B MK-8266 0.4 mg fasted and Panel B MK-8266 0.4 mg fed were combined in the analysis. One participant in Panel B 1.2 mg + 0.6 mg did not receive the 1.2 mg dose and was not included in this analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of central pulse pressure
Groups:
- Panel A Placebo; Panel B Placebo; Panel C Placebo: Placebo to MK-8266
- Pooled Panel B MK-8266 0.4 mg (Healthy Males): MK- 8266 single dose 0.4 mg in healthy male participants, fasted and fed
- Panel B MK-8266 1.2 mg (Healthy Males): MK-8266 single dose 1.2 mg in healthy male participants
- Panel B MK-8266 1.2/0.6 mg (Healthy Males): MK-826 6 single 1.2 mg followed in 6 hours by a 0.6 mg dose in healthy male participants
- Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod.: MK-8266 single 1.0 mg dose followed in 6 hours by a 0.6 mg dose followed in 6 hours by a 0.6 mg dose in participants with mild/mod. hypertension
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel A Placebo | Pooled Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B Placebo | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) | Panel C Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 6 | 5 | 8 | 6 | 6 | 6 | 6 | 12
Percentage of central pulse pressure | -8.79 (9.66) | -2.96 (9.15) | -1.73 (4.49) | -7.42 (3.85) | -5.70 (7.57) | -1.73 (7.36) | -13.1 (8.71) | -14.1 (7.49) | -16.7 (5.21) | -15.3 (2.68) | 8.43 (4.98) | 11.29 (6.60) | 7.78 (11.10) | 8.74 (3.90) | 17.74 (6.75)
Statistical Analysis 1: Comparison: Panel A MK-8266 0.1 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.003, ANOVA; 0.1 mg vs. placebo = -7.06, 90% CI 2-sided [-11.1 to -3.00]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.2 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.310, ANOVA; 0.2 mg vs. placebo = -1.23, 90% CI 2-sided [-5.42 to 2.96]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.5 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.498, ANOVA; 0.5 mg vs. placebo = 0.01, 90% CI 2-sided [-4.05 to 4.06]
Statistical Analysis 4: Comparison: Panel A MK-8266 1.0 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.012, ANOVA; 1 mg vs. placebo = -5.69, 90% CI 2-sided [-9.74 to -1.63]
Statistical Analysis 5: Comparison: Panel A MK-8266 1.0/0.8 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.059, ANOVA; 1 mg + 0.8 mg vs. placebo = -3.97, 90% CI 2-sided [-8.16 to 0.22]
Statistical Analysis 6: Comparison: Pooled Panel B MK-8266 0.4 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.191, ANOVA; 0.4 mg vs. placebo = 2.22, 90% CI 2-sided [-2.09 to 6.54]
Statistical Analysis 7: Comparison: Panel B MK-8266 1.2 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.333, ANOVA; 1.2 mg vs. placebo = 1.24, 90% CI 2-sided [-3.67 to 6.15]
Statistical Analysis 8: Comparison: Panel B MK-8266 1.2/0.6 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.314, ANOVA; 1.2 mg + 0.6 mg vs. placebo = -1.43, 90% CI 2-sided [-6.50 to 3.63]
Statistical Analysis 9: Comparison: Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.001, ANOVA; 1 mg + 0.8 mg vs. placebo = -9.31, 90% CI 2-sided [-14.2 to -4.37]
Statistical Analysis 10: Comparison: Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.017, ANOVA; 1.2 mg + 1.0 mg vs. placebo = -6.45, 90% CI 2-sided [-11.4 to -1.51]
Statistical Analysis 11: Comparison: Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. vs Panel C Placebo; Test type: Other; p = 0.001, ANOVA; 1.0 mg + 0.6 mg + 0.6 mg vs. placebo = -9.96, 90% CI 2-sided [-14.9 to -5.02]
Statistical Analysis 12: Comparison: Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.002, ANOVA; 1 mg + 1 mg + 0.6 mg vs. placebo = -9.00, 95% CI 2-sided [-13.8 to -4.17]

4. Primary Outcome: MK-8266 Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC[0-inf] is a measure of the mean concentration levels of drug in the plasma after the dose. AUC[0-inf] was not collected, analyzed or summarized for participants receiving placebo.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours postdose
Population: AUC[0-inf] was not estimated at MK-8266 doses <1.0 mg and for the first 2 doses in Panel C due to the lack of measureable concentrations, and for participants receiving placebo. One participant in Panel B 1.2 mg + 0.6 mg did not receive the 1.2 mg dose and was not included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/mL*hr
Groups:
- Panel A MK-8266 0.1 mg (Healthy Males): MK-826 6 single 0.1 mg dose in healthy male participants
- Panel A MK-8266 0.2 mg (Healthy Males): MK-826 6 single 0.2 mg dose in healthy male participants
- Panel A MK-8266 0.5 mg (Healthy Males): MK-826 6 single 0.5 mg dose in healthy male participants
- Panel A MK-8266 1.0 mg (Healthy Males): MK-826 6 single 1.0 mg dose in healthy male participants
- Panel A MK-8266 1.0/0.8 mg (Healthy Males): MK-826 6 single 1.0 mg dose followed in 6 hours by a 0.8 mg dose in healthy male participants
- Panel C MK- 8266 1.0/0.8 mg (Mild/Mod. Hypertension): MK-8266 single 1.0 mg dose followed in 8 hours by a 0.8 mg dose in participants with mild/mod. hypertension
- Panel C MK- 8266 1.2/1.0 mg (Mild/Mod. Hypertension): MK-8266 single 1.2 mg dose followed in 8 hours by a 1.0 mg dose in participants with mild/mod. hypertension
- Panel C MK- 8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension): MK-8266 single 1.0 mg dose followed in 6 hours by a 1.0 mg dose followed in 6 hours by a 0.6 mg dose in participants with mild/mod. hypertension
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK- 8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension)
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 0 | 6 | 5 | 0 | 0 | 0 | 6 | 6
mg/mL*hr |  |  |  | 264 (64.4) | 441 (105) |  | 216 (55.95) | 350 (49.5) |  |  |  | 528 (151) | 623 (350)

5. Primary Outcome: MK-8266 PK Parameter Observed Maximum (Peak) Plasma Concentration (Cmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. For Panel A 1.0/0.8 mg MK-8266, the second dose was not well characterized due to limited sampling. Observed exposure likely underestimates the true exposure. Cmax was not collected, analyzed or summarized for participants receiving placebo.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that their data likely exhibited the effects of treatment, according to the underlying scientific model. Cmax was not estimated for participants receiving placebo. One participant in Panel B 1.2 mg + 0.6 mg did not receive the 1.2 mg dose and was not included in this analysis.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK- 8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
nM | 2.28 (0.291) | 4.33 (0.454) | 11.4 (0.819) | 22.2 (3.40) | 20.5 (2.58) | 7.46 (1.41) | 19.5 (5.14) | 21.3 (4.16) | 7.71 (2.64) | 19.1 (3.77) | 22.1 (3.06) | 21.7 (3.80) | 22.4 (3.59)

6. Primary Outcome: MK-8266 PK Parameter Observed Time to Reach Cmax (Tmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. Tmax was not collected, analyzed or summarized for participants receiving placebo.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours postdose
Population: The analysis population consisted of participants who complied with the protocol sufficiently to ensure that their data likely exhibited the effects of treatment. Tmax was not estimated for participants receiving placebo. One participant in Panel B 1.2 mg + 0.6 mg did not receive the 1.2 mg dose and was not included in this analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK- 8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
Hours | 2.5 [1.5 to 4.0] | 4.0 [3.0 to 4.0] | 3.5 [2.0 to 4.0] | 4.0 [3.0 to 4.0] | 3.5 [2.0 to 8.0] | 3.0 [2.0 to 4.0] | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 4.0] | 1.5 [1.5 to 6.0] | 3.0 [2.0 to 10.0] | 5.0 [3.0 to 10.0] | 6.5 [2.0 to 15.0] | 9.0 [3.0 to 15.0]

7. Primary Outcome: MK-8266 PK Parameter Apparent t1/2
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. t1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. Harmonic means +/- Pseudo standard deviations are displayed. t1/2 was not collected, analyzed or summarized for participants receiving placebo.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours postdose
Population: t1/2 was not estimated at MK-8266 doses below 1 mg and for the first 2 doses in Panel C due to the lack of measureable concentrations and for participants receiving placebo. One participant in Panel B 1.2 mg + 0.6 mg did not receive the 1.2 mg dose and was not included in this analysis.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK- 8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK- 8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension)
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 0 | 6 | 5 | 0 | 0 | 0 | 6 | 6
Hours |  |  |  | 13.6 (2.6) | 11.7 (2.2) |  | 9.2 (3.5) | 12.0 (3.0) |  |  |  | 10.4 (2.2) | 12.8 (4.8)

8. Secondary Outcome: Effect of Food on MK-8266 PK Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24hr) Following Administration of Single Oral Doses of MK-8266 at 0.4 mg to Healthy Male Participants
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC[0-24 hours] is a measure of the mean concentration levels of drug in the plasma after the dose. The Fed Group was administered a high fat meal.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 postdose
Population: All participants who complied with the protocol sufficiently to ensure that their data likely exhibited the effects of treatment, according to the underlying scientific model.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM·hr
Arm/Group | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males)
Number analyzed (Participants) | 6 | 6
nM·hr | 59.6 [38.9 to 91.2] | 52.9 [34.6 to 81.0]
Statistical Analysis 1: Comparison: Panel B MK-8266 0.4 mg (Healthy Males) vs Panel B MK-8266 0.4 mg Fed (Healthy Males); Test type: Other; GMR (Fed/Fasted) = 0.89, 95% CI 2-sided [0.86 to 0.92]

9. Secondary Outcome: Effect of Food on MK-8266 PK Parameter Cmax Following Administration of Single Oral Doses of MK-8266 at 0.4 mg to Healthy Male Participants
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. The Fed Group was administered a high fat meal.
Time Frame: Predose, 0.5, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours postdose
Population: as for outcome 8
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males)
Number analyzed (Participants) | 6 | 6
nM | 7.5 [5.2 to 11.0] | 7.3 [5.0 to 10.6]
Statistical Analysis 1: Comparison: Panel B MK-8266 0.4 mg (Healthy Males) vs Panel B MK-8266 0.4 mg Fed (Healthy Males); Test type: Other; GMR (Fed/fasted) = 0.97, 95% CI 2-sided [0.79 to 1.19]

10. Secondary Outcome: Time-Weighted Average of Heart Rate (0-12 Hours)
Description: HR was measured with a validated automatic measuring device. Time weighted average was obtained as follows: For all HR values obtained over the 12-hour observation period, multiply the length of time that the participant spent at each HR value by that HR value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified HR value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Participants in Arms/Groups in which MK-8266 or placebo was administered in more than one period were counted separately for each period.
Time Frame: Up to 12 hours
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Beats per Minute
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel A Placebo | Pooled Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B Placebo | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) | Panel C Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 6 | 5 | 8 | 6 | 6 | 6 | 6 | 12
Beats per Minute | 58.79 (6.71) | 61.65 (3.06) | 56.36 (4.86) | 66.40 (7.90) | 63.71 (3.17) | 59.32 (6.28) | 57.38 (5.92) | 61.07 (5.04) | 59.92 (10.23) | 56.53 (6.66) | 69.82 (8.09) | 66.40 (9.82) | 64.14 (7.40) | 64.90 (8.33) | 60.66 (8.07)
Statistical Analysis 1: Comparison: Panel A MK-8266 0.1 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.396, ANOVA; 0.1 mg vs placebo = -0.53, 90% CI 2-sided [-3.92 to 2.86]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.2 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.1329, ANOVA; 0.2 mg vs. placebo = 2.33, 90% CI 2-sided [-1.17 to 5.83]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.5 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.0741, ANOVA; 0.5mg vs. placebo = -2.96, 90% CI 2-sided [-6.35 to 0.43]
Statistical Analysis 4: Comparison: Panel A MK-8266 1.0 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p < 0.001, ANOVA; 1 mg vs. placebo = 7.08, 90% CI 2-sided [3.69 to 10.47]
Statistical Analysis 5: Comparison: Panel A MK-8266 1.0/0.8 mg (Healthy Males) vs Panel A Placebo; Test type: Other; p = 0.0211, ANOVA; 1 mg + 0.8 mg vs. placebo = 4.39, 90% CI 2-sided [0.89 to 7.09]
Statistical Analysis 6: Comparison: Pooled Panel B MK-8266 0.4 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.399, ANOVA; 0.4 mg vs. placebo = 0.85, 90% CI 2-sided [-4.79 to 6.48]
Statistical Analysis 7: Comparison: Panel B MK-8266 1.2 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.100, ANOVA; 1.2 mg vs. placebo = 4.54, 90% CI 2-sided [-1.94 to 11.02]
Statistical Analysis 8: Comparison: Panel B MK-8266 1.2/0.6 mg (Healthy Males) vs Panel B Placebo; Test type: Other; p = 0.195, ANOVA; 1.2 mg + 0.6 mg vs. placebo = 3.38, 90% CI 2-sided [-3.29 to 10.06]
Statistical Analysis 9: Comparison: Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.022, ANOVA; 1.0 mg + 0.8 mg vs. placebo = 9.16, 90% CI 2-sided [1.74 to 16.58]
Statistical Analysis 10: Comparison: Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.098, ANOVA; 1.2 mg + 1.0 mg vs. placebo = 5.74, 90% CI 2-sided [-1.68 to 13.16]
Statistical Analysis 11: Comparison: Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. vs Panel C Placebo; Test type: Other; p = 0.214, ANOVA; 1 mg + 0.6 mg + 0.6 mg vs. placebo = 3.48, 90% CI 2-sided [-3.94 to 10.90]
Statistical Analysis 12: Comparison: Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) vs Panel C Placebo; Test type: Other; p = 0.163, ANOVA; 1 mg + 1 mg + 0.6 mg vs. placebo = 4.24, 95% CI 2-sided [-3.03 to 11.52]

ADVERSE EVENTS:
Time Frame: Up to 14 days after administration of the last dose of study drug (Up to 43 days)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The analysis population consisted of all participants who received at least one dose of the investigational drug.
Groups:
- Panel B MK-8266 1.2/0.6 mg (Healthy Males): MK-8266 single 1.2 mg followed in 6 hours by a 0.6 mg dose in healthy male participants
Arm/Group | Panel A MK-8266 0.1 mg (Healthy Males) | Panel A MK-8266 0.2 mg (Healthy Males) | Panel A MK-8266 0.5 mg (Healthy Males) | Panel A MK-8266 1.0 mg (Healthy Males) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) | Panel B MK-8266 0.4 mg (Healthy Males) | Panel B MK-8266 1.2 mg (Healthy Males) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) | Panel B MK-8266 0.4 mg Fed (Healthy Males) | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) | Pooled Placebo (Panels A, B, C)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/23
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 5/6 | 2/6 | 3/6 | 1/6 | 4/6 | 3/6 | 2/6 | 3/6 | 4/6 | 6/6 | 3/6 | 10/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A MK-8266 0.1 mg (Healthy Males) (N=6) | Panel A MK-8266 0.2 mg (Healthy Males) (N=6) | Panel A MK-8266 0.5 mg (Healthy Males) (N=6) | Panel A MK-8266 1.0 mg (Healthy Males) (N=6) | Panel A MK-8266 1.0/0.8 mg (Healthy Males) (N=6) | Panel B MK-8266 0.4 mg (Healthy Males) (N=6) | Panel B MK-8266 1.2 mg (Healthy Males) (N=6) | Panel B MK-8266 1.2/0.6 mg (Healthy Males) (N=6) | Panel B MK-8266 0.4 mg Fed (Healthy Males) (N=6) | Panel C MK-8266 1.0/0.8 mg (Mild/Mod. Hypertension) (N=6) | Panel C MK-8266 1.2/1.0 mg (Mild/Mod. Hypertension) (N=6) | Panel C MK-8266 1.0/0.6/0.6 mg (Mild/Mod. Hypertension) (N=6) | Panel C MK-8266 1.0/1.0/0.6 mg (Mild/Mod. Hypertension) (N=6) | Pooled Placebo (Panels A, B, C) (N=23)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 5 (8) | 3 (3) | 6 (9)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.